CLINICAL TRIAL: NCT04677075
Title: New Formula to Predict Failure of Primary Closure and the Need for Reconstructive Coverage Following Mastectomy.
Brief Title: New Formula to Predict the Need for Reconstructive Coverage Following Mastectomy
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Joseph Rizk Awad, lecturer of surgery, Zagazig University
Other Study IDs: mastectomy coverage formula 20
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Neoplasms
Keywords: post mastectomy coverage, raw area
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mastectomy group: patients with breast cancer and eligible for mastectomy
  Interventions: Procedure: mastectomy

INTERVENTIONS:
Procedure: mastectomy — mastectomy either simple or modified radical

SUMMARY:
Mastectomy is a cornerstone operative procedure in breast cancer treatment leaving a raw area behind with possibility of failure of primary closure sometimes with unavailability of facilities of reconstruction. This opened the door for this research to find a formula to predict the need of reconstruction

DETAILED DESCRIPTION:
Surgical intervention for breast cancer includes dealing with the primary tumour, added to it is the axillary dissection with variable options in both of them according to multiple factors. Mastectomy represents a part of several operations as radical and modified radical mastectomy, while in others it may be the whole operation as in palliative simple mastectomy. Moreover, re-excision of local recurrence is another form of surgical intervention.

At the step of mastectomy or re-excision of locally recurrent disease, the challenge of closure may arise, as simple primary closure may not be possible because of wide wound gap. In this situation, reconstruction is unavoidably needed and this situation represents one of two situations in which reconstruction is indicated.

As reconstruction sometimes needs certain expertise which may not be available momentarily and needs previous arrangement. Moreover sometimes mastectomy exceeds the previous expectation leaving a big gap beyond simple approximation, so the investigators developed a formula to assess the need of reconstructive coverage.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer primary or recurrent, early, locally advanced or metastatic, as long as they were assigned to be treated with any procedure in which mastectomy is part or all of the procedure, were included in this study.

Exclusion Criteria:

1. Any patient diagnosed with breast cancer and planned to be treated with conservative breast cancer
2. Any patient whose design for excision was not regular ellipse but an irregularly tailored excision margin
3. Any patient with ischemic flaps (due to excessive tension or wrong dissection) following mastectomy
4. Any patient had skin disease affecting its healthiness

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: breast care clinic
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Clavicle-7th rib/sternal length ratio | for each patient at time of operation
  the ratio of clavicle-7th rib in relation to the length of the sternum
Upper flap length stretch ratio | for each patient at time of operation
  the ratio of the perpendicular line from the highest point of the upper border of mastectomy ellipse to the clavicle originally in relation to the length after stretch
Lower flap length stretch ratio | for each patient at time of operation
  the ratio of the perpendicular line from the lowest point of the lower border of mastectomy ellipse to the 7th rib originally to the length after stretch

SECONDARY OUTCOMES:
flap index | through study completion, an average of 3 years
  entangling of the above measurement in an equation to yield a number so when the distance from the clavicle to the 7th rib (in the midclavicular plane) is subtracted from it, a number is yielded, predicting the feasibility of closure without need to reconstruction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Zagazig, Sharqia Province, Egypt